CLINICAL TRIAL: NCT02758795
Title: Antiinflammatory Effect of Dietary Protein Intake in Elderly People
Acronym: AEDP
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Limerick (Other)
Collaborators: Ireland: Department Agriculture Food and the Marine (Unknown)
Responsible Party: Principal Investigator, Phil Jakeman, Professor, University of Limerick
Allocation: Randomized | Model: Crossover | Masking: Single | Purpose: Basic Science
Other Study IDs: FIRM2016
Record Dates: First submitted 2016-02-12; First posted 2016-05-03 (Estimated); Last update posted 2017-08-01 (Actual); Status verified 2017-07

CONDITIONS: Inflammation
Keywords: protein; inflammation; anti-inflammatory agents
MeSH Terms: conditions — Inflammation | interventions — Nutrients

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- CONTROL (Placebo Comparator): A placebo nutrient drink with no anti-inflammatory bioactivity (measure by cell bioassay in vitro) Dose provided per kg of body mass: 0.33g protein mixed in 500ml of water as a protein 'shake' Energy ~ 160 kcal
  Interventions: Dietary Supplement: CONTROL
- NUTRIENT (Active Comparator): A nutrient drink with confirmed anti-inflammatory bioactivity (measured by cell bioassay in vitro) Dose provided per kg of body mass: 0.33g protein mixed in 500ml of water as a protein 'shake' Energy ~ 160 kcal
  Interventions: Dietary Supplement: NUTRIENT

INTERVENTIONS:
Dietary Supplement: CONTROL — Following an overnight fast, participants submit to cannulation of a superficial arm vein from which are drawn serial samples of blood prior to and for 3 hours following ingestion of a prescribed protein 'shake'
  Arms: CONTROL
Dietary Supplement: NUTRIENT — Following an overnight fast, participants submit to cannulation of a superficial arm vein from which are drawn serial samples of blood prior to and for 3 hours following ingestion of a prescribed protein 'shake'
  Arms: NUTRIENT

SUMMARY:
The aim is to evaluate the effect of ingestion of a modified bovine milk protein on circulating markers of inflammation in healthy men and women aged 50-70y.The focus is healthy ageing, i.e. delaying the deterioration in health status in older adults. Loss of lean tissue mass, termed sarcopenia is a consequence of aging per se, modified by nutrition and lifestyle behaviour. Advancing the prospect of 'successful aging' a 6-month period of protein-based nutritional support has shown preservation/accrual of lean tissue. Chronic low-grade inflammation is common in ageing and is a compounding factor leading to 'anabolic blunting', i.e. a reduced sensitivity of lean tissue to enhance the synthesis of lean tissue mass in response to protein feeding. Using a simulated human gastrointestinal digestion model we have recently shown proteins to have an anti-inflammatory bioactivity in vitro. This study investigates whether the anti-inflammatory response is retained, post-digestion in vivo.

DETAILED DESCRIPTION:
Participants to be recruited, are aged 50 to 70y from the Healthy Aging Study (EHSREC10_45) who will attend on 4 test days (occasions)

Study Design: Single blind, randomised, repeated measures design with 2 independent factor (time x treatment)

Procedures:

Occasion 1 Subjects will undertake a preliminary assessment as per EHSREC 10_45 as follows; i. medical history and examination by a qualified medical doctor (~45 min); ii. provide a blood and urine sample to be evaluated (following analysis) by a qualified medical doctor;

Occasion 2 Subjects will then undertake, as per EHSREC 2013 01_12, an assessment of body composition, dietary intake and habitual physical activity as follows; iii. habitual food intake evaluated by a qualified dietitian (~45 min); iv. body composition (~45 min) v. habitual physical activity level (PAL) quantified using the European Physical Activity Questionnaire (EPAQ-2; ~ 15 min).

Occasion 3/4

Subjects will then undertake two controlled feeding trials, each trial separated by approximately 7 days as follows:

Subjects will report to the Metabolic Laboratory (PG-052b), Physical Education and Sports Sciences (PESS) Building following an overnight fast.

(i) A cannula will be inserted into a peripheral arm vein by a qualified clinician or phlebotomist;

(ii) a 10ml blood sample will be withdrawn and aliquots generated for subsequent analysis; (iii) Following a 15 min rest period subjects will be given in randomised order either control (CONTROL) - a placebo nutrient drink (per kg of body mass: 0.33g protein with no anti-inflammatory bioactivity; energy ~ 160 kcal in 500ml water) or nutrient (NUTRIENT) - a nutrient drink (per kg of body mass: 0.33g protein with confirmed anti-inflammatory bioactivity; energy ~ 160 kcal in 500ml water) to be consumed within a 10 minute period.

CONTROL and NUTRIENT will be reversed for the 2nd trial in randomised order.

(iv) Whilst remaining sitting at rest (reading, undertaking computer work etc.) further blood samples will be withdrawn at 0, 15, 30, 45, 60 75, 90, 120 and 180 minutes post feeding.

Total blood draw = 100ml per trial.

Data Analysis: (i) Shapiro-Wilk test of normality, then (ii) repeated measures analysis either by ANOVA(R) if normal or Friedman Test if non-normally distributed.

ELIGIBILITY:
Inclusion Criteria:

* Men and Women
* Aged 50 to 70y
* Conducted by a medical doctor and based on Grieg et al. 1994 to be 'healthy' (i.e. 'disease-free') free-living and fully mobile

Exclusion Criteria:

* Age <50 or > 70y.
* Contraindication identified by medical doctor based on Grieg et al. 1994 definition of 'healthy' (i.e. 'disease-free') free-living and fully mobile older subjects
* Lactose intolerant or intolerance to dairy-based foods.

Ages: 50 Years to 70 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 16 (Actual)
Dates: Start 2016-02; Primary Completion 2017-04-08 (Actual); Study Completion 2017-04-08 (Actual)

PRIMARY OUTCOMES:
Interleukin 6 (IL-6) response of macrophage cells to stimulation with bacterial lipopolysaccharide (LPS) | All timepoints to 180 min following ingestion of NUTRIENT and CONTROL drinks
  Macrophages seeded at a density of 0.2 x 10^5 cells/ml, stimulated with LPS (0.1ug/ml) and incubated for 24h in serum obtained from subjects reported as %of control value, i.e. relative to cells incubated without human serum
Tumour necrosis factor alpha (TNF-alpha) response of macrophage cells to stimulation with bacterial lipopolysaccharide (LPS) | All timepoints to 180 min following ingestion of NUTRIENT and CONTROL drinks
  Macrophages seeded at a density of 0.2 x 10^5 cells/ml, stimulated with LPS (0.1ug/ml) and incubated for 24h in serum obtained from subjects reported as %of control value, i.e. relative to cells incubated without human serum
Interleukin-1 beta (IL1_beta) response of macrophage cells to stimulation with bacterial lipopolysaccharide (LPS) | All timepoints to 180 min following ingestion of NUTRIENT and CONTROL drinks
  Macrophages seeded at a density of 2 x 10^5 cells/ml, stimulated with LPS (0.2ug/ml) and incubated for 24h in serum obtained from subjects reported as %of control value, i.e. relative to cells incubated without human serum

CONTACTS AND LOCATIONS:
Overall Officials: Philip Jakeman, PhD, Principal Investigator — University of Limerick
Locations (1):
- University of Limerick, Limerick, Co Limerick, Ireland